CLINICAL TRIAL: NCT06104267
Title: A Single-Arm, Prospective, Exploratory Study to Evaluate Feasibility and Effect of Medical Tai Chi Exercise Healing in Treating mCRC Patients
Brief Title: Medical Tai Chi Exercise Healing in Treating mCRC Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: SIR RUNRUN Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KEEP-G 10
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical Tai Chi Exercise Group (Experimental)
  Interventions: Behavioral: 7-Form of Medical Tai Chi Exercise Healing for Colon cancer patients

INTERVENTIONS:
Behavioral: 7-Form of Medical Tai Chi Exercise Healing for Colon cancer patients — The programme is based on the "7-Form of Medical Tai Chi Exercise Healing for Colon cancer patients" that lasted 60 minutes three times a week for eight weeks and is led by a Tai Chi instructor with more than 5 years of teaching experience. Each session included a warm-up, movement instruction, breathing techniques, and relaxation. To ensure that each participant is proficient in Tai Chi, they will take at least 2 sessions of 60-minute Tai Chi training before the start of the intervention, until they are able to perform all Tai Chi movements correctly and successfully, and record a video to be used in software for practice at home. The enrolled patients, Tai Chi instructors and relevant staff of the subject group set up a WeChat group, and the enrolled patients, outside of the prescribed practice time each week, can practice at home or outdoors by themselves. They can send the video of the practice to the WeChat group.

SUMMARY:
As a traditional martial art in China, Tai Chi Chuan has excellent health benefits along with its combat function.Studies have shown that Tai Chi as an exercise prescription can significantly reduce the incidence of cancer, but the complexity of Tai Chi Chuan routines, poor disease targeting, and the lack of traditional internal mental and physical training method limit the healing of tumours and other diseases. For this reason, we have established the Medical Tai Chi Exercise Healing System（MTCEH）, which integrates Tai Chi exercise, traditional Chinese internal mental and physical training method, rehabilitation medicine and sports medicine methods, on the basis of evidence-based medicine and with the aim of targeting different tumour treatments. With the characteristics of easily learning, internal and external training, and individualised treatment of tumours, this series of routines effectively combines traditional oriental Tai Chi martial arts with tumour treatment, which opens up a beautiful and mysterious oriental healing journey for integrative medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological documentation of adenocarcinoma of the colon or rectum.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
3. Life expectancy of at least 6 months.
4. Adequate bone marrow, liver, cardiac and renal function as assessed by the laboratory required by protocol（ALT/AST≤2.5×UNL or ≤5×UNL with liver metastasis,TBIL≤2.5×UNL,Cr≤1.5×UNL,WBC≥3×109/L,NE≥1.5×109/L，PLT≥80×109/L，Hb≥90g/L,PT-INR/APTT <1.5UNL; LVEF≥ 50%）.
5. Subjects must complete the treatment and follow-up on schedule according to the research plan.

Exclusion Criteria:

1. Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
2. Any serious or unstable medical condition、mental illness or known active alcohol or drug abuse or dependence.
3. Unhealed surgical wounds and intolerance
4. Extreme fatigue, anemia (<80 g/L) or dystaxia
5. toxicity grade ≥III in chemoradiotherapy or targeted therapy (NCI-CTCAE 5.0), or severe intolerance
6. exercise contraindications for patients with cardiovascular diseases or pulmonary diseases (referring to the Chinese Guideline for Cardiac Rehabilitation and Secondary Prevention [edition 2018] and Evidence-based Practice Guidelines for Clinical Rehabilitation of Chronic obstructive Pulmonary Disease [edition 2021]); uncontrolled unstable angina, diastolic dysfunction grade IV, uncontrolled severe arrhythmia, uncontrolled hypertension;
7. high fever, serious infection, dyscrasia, multiple organ failure, or incapability to cooperate
8. thrombosis in the active phase
9. For female subjects: they should be surgical sterilized, postmenopausal patients, or agree to use a medically approved contraceptive method during the study treatment period and within 6 months after the end of the study treatment period; The serum or urine pregnancy test must be negative within 7 days before enrollment and must be non lactating. Male subjects: patients who agree to use a medically approved contraceptive method during the study treatment period and within 6 months after the end of the study treatment period.
10. other conditions confirmed by the multidisciplinary cancer rehabilitation team.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence rates | post 8-week intervention
  The adherence rates will be measured by the number of tai chi sessions performed divided by the total possible tai chi sessions

SECONDARY OUTCOMES:
the Brief Fatigue Inventory (BFI) | post 8-week intervention
the Pittsburgh Sleep Quality Index (PSQI) | post 8-week intervention
EORTC - Quality of Life | post 8-week intervention
self-rating anxiety scale（SAS） | post 8-week intervention
self-rating depression scale（SDS） | post 8-week intervention

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided